CLINICAL TRIAL: NCT02429050
Title: Morphine for Palliative Treatment of Refractory Dyspnea in Patients With Advanced COPD: Benefits and Respiratory Adverse Effects
Brief Title: Morphine for Treatment of Dyspnea in Patients With COPD
Acronym: MORDYC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 152002; 80-83600-98-3006 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2015-04-02; First posted 2015-04-29 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Dyspnea; Breathlessness; Morphine; Opioid; Symptom Management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): sustained release morphine
  Interventions: Drug: sustained release morphine
- control (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sustained release morphine — Patients will receive morphine SR 10mg two to three times daily or placebo. Hard gelatin capsules of size AA in Swedish orange containing one morphine SR tablet 10 mg per capsule will be produced. Morphine SR has a marketing authorisation for pain and will be used according to current Dutch and international guidelines for treatment of dyspnea.
  Arms: intervention
Drug: placebo — Patients in the control group will receive placebo, consisting of microcrystalline cellulose (FMC BioPolymer). Hard gelatin capsules of size AA in Swedish orange containing microcrystalline cellulose will be produced.
  Arms: control

SUMMARY:
Dyspnea is the most reported symptom of patients with advanced Chronic Obstructive Pulmonary Disease (COPD) and is undertreated. Morphine is an effective treatment for dyspnea and is recommended in clinical practice guidelines, but questions concerning benefits and concerns about respiratory adverse effects remain. For example, the effect on health-related quality of life and functional capacity is unknown. In one-third of the patients oral sustained release morphine (morphine SR) doesn't relieve dyspnea and it remains unknown whether severity and descriptors of breathlessness may predict a response to morphine. Finally, cost-effectiveness of morphine SR in this patient group is unknown. Therefore, prescription of morphine to patients with COPD is limited.

Objectives of this double blind randomized controlled trial are to study the effect of oral administration of morphine SR on health-related quality of life, respiratory adverse effects, and functional capacity; to explore whether description and severity of breathlessness are related with a clinically relevant response to morphine and to analyse the cost-effectiveness of morphine SR. The study population will consist of 124 clinically stable outpatients with COPD and severe dyspnea despite optimal pharmacological and non-pharmacological treatment.

DETAILED DESCRIPTION:
Participants will be outpatients with a confirmed diagnosis of COPD, who suffer from severe dyspnea despite optimal pharmacological and non-pharmacological treatment. Participants will be recruited at CIRO, a center for pulmonary rehabilitation in the Netherlands after they completed a pulmonary rehabilitation program. After providing informed consent, patients will be randomized. Members of the research team who perform measurements will be blinded for treatment allocation.

Patients in the intervention group will receive regular clinical care and morphine SR 10mg, administered twice daily (20mg/24h), which can be increased after one or two weeks to three times per day 10mg (30mg/24h) in non-responders. Patients will be defined as non-responders if the mean dyspnea numeric rating scale (NRS) score was not reduced by 1 point in comparison with baseline. The control group will receive regular clinical care and placebo medication. Patients will receive morphine or placebo for four weeks. In addition, both groups will receive a prescription for a laxative and metoclopramide at the start of the intervention and will be instructed to adjust the dose as needed.

When the intervention period has ended, participants can choose to continue morphine treatment. They will be followed for twelve weeks to assess their healthcare use, use of morphine and number of adverse effects and exacerbations.

Measurements at baseline will include: demographics, medical history, medication, co-morbidities, exercise capacity, respiratory parameters, generic and disease-specific health-related quality of life (HRQoL), severity of dyspnea, sensory and affective dimensions of dyspnea, impact of dyspnea, cognition, level of daytime sleepiness, and functional capacity. A member of the research team will visit patients after 1 and 2 weeks in their home environment to assess adverse effects, compliance, exacerbations, disease-specific HRQoL, mobility, severity of dyspnea, and some respiratory parameters. A member of the research team will call the patient after 2 days and 3 weeks to assess adverse effects, compliance, exacerbations, and severity of dyspnea. After 4 weeks the following measurements will be performed: respiratory parameters, exercise capacity, general and disease-specific HRQoL, sensory and affective dimensions of dyspnea, impact of dyspnea, functional capacity, and adverse effects. Overnight oximetry will be performed in the home environment at baseline and after four weeks. A diary for costs and healthcare use will be filled in during four weeks.

Measurements during the twelve weeks following the intervention include: retrospective cost questionnaire, generic and disease-specific quality of life severity of dyspnea and adverse effects.

Statistical analyses Baseline characteristics will be compared between the intervention and control group using descriptive statistics. Chi square tests will be used for categorical variables. Independent sample T-tests and Mann-Whitney U-tests will be used for continuous variables, according to the variable distribution. Change in CAT-score, respiratory parameters and 6MWD between baseline and four weeks will be compared between patients in the intervention and the control group. First, mean change in CAT-score, respiratory parameters and 6MWD will be compared between the two groups using an independent sample T-test or Mann-Whitney U test, according to the variable distribution. Afterwards, multivariate analyses for longitudinal data will be performed. Analyses will be done using an intention-to-treat approach. The relationship between response to opioids and severity of dyspnea and descriptors of breathlessness will be explored using univariate analysis, followed by a binary logistic regression model. A trial-based economic evaluation will be performed, based on empirical data obtained in the RCT. The economic evaluation will be performed from the societal and healthcare perspective, the first including costs inside and outside the health care sector, and will follow published international guidelines. The time horizon of the trial-based economic evaluation will be four weeks. The outcomes of the twelve weeks following the intervention will be used in the model-based economic evaluation. The model will probably take the form of a Markov model; however this will be decided upon during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to the current Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (GOLD);
* Optimal pharmacological treatment, including including treatment with a combination of a long-acting muscarinic antagonist and an ultra-long-acting β-agonist;
* Grade 3 or 4 dyspnea on the mMRC dyspnea scale;
* Optimal non-pharmacological treatment defined as completed a comprehensive pulmonary rehabilitation program.

Exclusion Criteria:

* History of substance misuse;
* Exacerbation of COPD within two weeks of study enrolment;
* Waiting list for lung transplantation;
* Pregnant or childbearing potential not using contraception;
* Renal failure (creatinine clearance <15mL/min);
* Not being able to read or fill in the questionnaires or diary;
* Allergy for morphine or its excipients;
* Concomitant use of irreversible MAO blockers;
* Use of opioids;
* History of convulsions;
* Head injury;
* Intestinal obstruction;
* Gastroparesis;
* Liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Disease-specific health-related quality of life (COPD Assessment Test (CAT)) | sixteen weeks
  Change in disease-specific health-related quality of life in four weeks measured with CAT
Change in partial pressure of CO2 (pCO2) | four weeks
  Change in pCO2 in four weeks
Change in partial pressure of O2 (pO2) | four weeks
  Change in pO2 in four weeks
Respiratory rate | four weeks
  Change in respiratory rate in four weeks
Pulse oximetric saturation (SpO2) | four weeks
  Change in SpO2 in four weeks
Transcutaneous carbon dioxide (PtcCO2) | four weeks
  Change in PtcCO2 in four weeks
Oxygen saturation during the night | four weeks
  Change in oxygen saturation during the night in four weeks using overnight oximetry

SECONDARY OUTCOMES:
distance walked in 6 Minute Walking Test (6-MWT) | four weeks
  Change in exercise capacity in four weeks measured with 6-MWT
Care dependency (Care Dependency Scale (CDS) | four weeks
  Change in care dependency in four weeks measured with CDS
Mobility (Timed 'Up & Go' (TUG) test) | four weeks
  Change in mobility in four weeks measured with TUG test.
Sensory and affective dimensions of dyspnea (Multidimensional Dyspnea Profile (MDP) | four weeks
  Sensory and affective dimensions of dyspnea in four weeks measured with MDP
Impact of dyspnea (Pulmonary Functional Status and Dyspnea Questionnaire, PFSDQ-M) | four weeks
  Change in impact of dyspnea in four weeks measured with PFSDQ-M
Severity of dyspnea (Numeric Rating Scale (NRS) | sixteen weeks
  Change in severity of dyspnea in four weeks measured with NRS
Daytime sleepiness (Epworth Sleep Questionnaire) | four weeks
  Change in level of daytime sleepiness in four weeks measured with Epworth Sleep Questionnaire
Cognition (Montreal Cognitive Assessment, (MoCA) | four weeks
  Change in cognition in four weeks measured with MoCA
Number of patients with adverse effects | sixteen weeks
  Adverse effects, including nausea, vomiting, constipation, drowsiness
Intake of medication | four weeks
  Number of missed medication intakes in four weeks
Number of exacerbations | sixteen weeks
  Number of exacerbations in four weeks
Cost of healthcare use in euro's | sixteen weeks
  Cost of healthcare use in euro's based on the number of hospitalizations, number and type of contact with physician, use of (professional) homecare, use of medication and absence of (voluntary) work due to illness

CONTACTS AND LOCATIONS:
Overall Officials: Daisy JA Janssen, MD, PhD, Principal Investigator — Maastricht UMC; E. FM Wouters, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Ciro centre of expertise for chronic organ failure, Horn, Netherlands

REFERENCES:
- [Derived] Verberkt CA, van den Beuken-van Everdingen MHJ, Dirksen CD, Schols JMGA, Wouters EFM, Janssen DJA. Cost-effectiveness of sustained-release morphine for refractory breathlessness in COPD: A randomized clinical trial. Respir Med. 2021 Apr;179:106330. doi: 10.1016/j.rmed.2021.106330. Epub 2021 Feb 10. PMID 33611087
- [Derived] Verberkt CA, van den Beuken-van Everdingen MHJ, Schols JMGA, Hameleers N, Wouters EFM, Janssen DJA. Effect of Sustained-Release Morphine for Refractory Breathlessness in Chronic Obstructive Pulmonary Disease on Health Status: A Randomized Clinical Trial. JAMA Intern Med. 2020 Oct 1;180(10):1306-1314. doi: 10.1001/jamainternmed.2020.3134. PMID 32804188